CLINICAL TRIAL: NCT07219550
Title: A Clinical Study to Evaluate the Effect of Hepatic Impairment on the Single-Dose Pharmacokinetics of MK-1084
Brief Title: A Study of MK-1084 in Participants With Hepatic Impairment and Healthy Volunteers (MK-1084-017)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1084-017; MK-1084-017 (Other: MSD)
Record Dates: First submitted 2025-10-20; First posted 2025-10-22 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Healthy; Hepatic Impairment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MK-1084 (Experimental): All participants will receive a single oral dose of MK-1084 on Day 1.
  Interventions: Drug: MK-1084

INTERVENTIONS:
Drug: MK-1084 — Oral Tablet

SUMMARY:
The purpose of this study is to learn what happens to MK-1084 levels in a person's body over time. Researchers will measure what happens to MK-1084 levels in the body when it is given to participants with hepatic (liver) impairment and healthy participants. Researchers also want to learn about the safety of MK-1084 when it is given to people with hepatic impairment and if people with hepatic impairment can tolerate it.

ELIGIBILITY:
The main inclusion criteria include but are not limited to:

All participants:

* Has a body mass index (BMI) between 18.0 and 42.0 kg/m^2

Participants with hepatic impairment (HI):

* Has a diagnosis of chronic, stable hepatic insufficiency at screening with features of cirrhosis

Healthy volunteers:

* Is medically healthy with no clinically significant medical history

The main exclusion criteria include but are not limited to:

All participants:

* Has a history of gastrointestinal disease which may affect food and drug absorption
* Has a history of cancer (malignancy)
* Has a positive result for human immunodeficiency virus (HIV)
* Has had major surgery and/or donated or lost significant volume of blood within 56 days prior to dosing

Participants with HI:

* Has had severe complications of liver disease within the preceding 3 months of screening
* Has a history of recent (within 3 months prior to screening) variceal bleeds
* Has evidence of hepatorenal syndrome
* Is not in sufficient health, with regard to stability of HI, to undergo participation in the study with anticipated survival of < 3 months
* Has a history of liver or other solid organ transplantation
* Has an active infection requiring systemic therapy
* Requires paracentesis more often than 2 times per month
* Has transjugular intrahepatic portosystemic shunt and/or has undergone portacaval shunting
* Has received antiviral and/or immune modulating therapy for hepatitis B virus (HBV) or hepatitis C virus (HCV) within 90 days prior to dosing
* Is using HIV protease inhibitors
* Is positive for Hepatitis B surface antigen (HBsAg)
* Is positive for HCV

Healthy volunteers:

* Has positive results for HBsAg or HCV

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Area Under the Concentration Versus Time Curve from 0 to the Time of the Last Quantifiable Sample (AUC0-last) of MK-1084 | At designated timepoints up to approximately 7 days post-dose
  Blood samples will be collected to determine the AUC0-last of MK-1084 in plasma.
Area Under the Concentration Versus Time Curve from 0 to Infinity (AUC0-inf) of MK-1084 | At designated timepoints up to approximately 7 days post-dose
  Blood samples will be collected to determine the AUC0-inf of MK-1084 in plasma.
Area Under the Concentration Versus Time Curve from 0 to 24 hours post-dose (AUC0-24) of MK-1084 | Up to approximately 24 hours post-dose
  Blood samples will be collected to determine the AUC0-24 of MK-1084 in plasma.
Maximum Observed Drug Concentration (Cmax) of MK-1084 | At designated timepoints up to approximately 7 days post-dose
  Blood samples will be collected to determine the Cmax of MK-1084 in plasma.
Time to Maximum Observed Drug Concentration (Tmax) of MK-1084 | At designated timepoints up to approximately 7 days post-dose
  Blood samples will be collected to determine the Tmax of MK-1084 in plasma.
Apparent Terminal Half-life (t1/2) of MK-1084 | At designated timepoints up to approximately 7 days post-dose
  Blood samples will be collected to determine the t1/2 of MK-1084 in plasma.
Apparent Clearance (CL/F) of MK-1084 | At designated timepoints up to approximately 7 days post-dose
  Blood samples will be collected to determine the CL/F of MK-1084 in plasma.
Apparent Volume of Distribution During Terminal Phase (Vz/F) of MK-1084 | At designated timepoints up to approximately 7 days post-dose
  Blood samples will be collected to determine the Vz/F of MK-1084 in plasma.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 14 days
  An AE is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. The number of participants experiencing AEs will be reported.
Number of Participants Who Discontinue Study Due to an AE | Up to approximately 14 days
  An AE is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. The number of participants discontinuing the study due to AEs will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (3):
- United States (3):
  - Arizona Clinical Trials ( Site 0003), Chandler, Arizona
  - Orlando Clinical Research Center ( Site 0001), Orlando, Florida
  - The Texas Liver Institute ( Site 0002), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/